CLINICAL TRIAL: NCT03312894
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-653 in the Treatment of Subjects With Treatment-Resistant Depression
Brief Title: Efficacy and Safety of TAK-653 in Treatment-Resistant Depression
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-653-2001; 2017-002232-16 (Registry Identifier: EudraCT); U1111-1200-8817 (Other: WHO); 17/SC/0606 (Registry Identifier: NRES); FAGG/R&D/LFT (Other: Federal Agency for Medicines and Health Products)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Treatment-Resistant Depression
Keywords: Drug therapy
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Ketamine Responders): TAK-653 6 mg (Experimental): TAK-653 tablets plus TAK-653 placebo-matching tablets, orally, once daily on Days 1 and 2; followed by TAK-653 tablets, orally, once daily on Days 3 and 4; followed by TAK-653 tablets plus TAK-653 placebo-matching tablets, orally, once daily on Days 5 to 7; followed by TAK-653 tablets, orally, once daily on Days 8 to 56.
  Interventions: Drug: TAK-653; Drug: Placebo
- Cohort 1 (Ketamine Responders): Placebo (Placebo Comparator): TAK-653 placebo-matching tablets, orally, once daily up to Day 56
  Interventions: Drug: Placebo
- Cohort 2 (Ketamine Nonresponders): TAK-653 6 mg (Experimental): TAK-653 tablets plus TAK-653 placebo-matching tablets, orally, once daily on Days 1 and 2; followed by TAK-653 tablets, orally, once daily on Days 3 and 4; followed by TAK-653 tablets plus TAK-653 placebo-matching tablets, orally, once daily on Days 5 to 7; followed by TAK-653 tablets, orally, once daily on Days 8 to 56.
  Interventions: Drug: TAK-653; Drug: Placebo
- Cohort 2 (Ketamine Nonresponders): Placebo (Placebo Comparator): TAK-653 Placebo-matching tablets, orally, once daily up to Day 56
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAK-653 — TAK-653 tablets
  Arms: Cohort 1 (Ketamine Responders): TAK-653 6 mg; Cohort 2 (Ketamine Nonresponders): TAK-653 6 mg
Drug: Placebo — Placebo-matching tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy of TAK-653 compared with placebo in maintaining the effect of ketamine treatment on depressive symptoms.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-653. TAK-653 is being tested to treat people who have depression and have not responded to several treatments (treatment-resistant depression).

This study will look at the efficacy and safety of TAK-653 in participants with treatment-resistant depression who take TAK-653 in addition to standard care.

The study will enroll approximately 90 patients. Participants who meet the study entry criteria will be assessed for response to ketamine by administering 2 intravenous (IV) infusions of ketamine (0.5 mg/kg given over 40 minutes; maximum dose 40 mg/day) on Day -5 (±1) and Day -1 (±1). To determine response to ketamine, the Day -5 predose Montgomery Åsberg Depression Rating Scale (MADRS) total score (before the first ketamine infusion) will be compared with the MADRS total score predose on Day 1 (24 hours after the second ketamine infusion on Day -1). Two cohorts (ketamine responders and ketamine nonresponders) of participants will be enrolled in parallel into the study.

Participants will then be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups - which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-653
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take one tablet at the same time each day throughout the study. This multi-center trial will be conducted worldwide. The overall time to participate in this study is 78 days. Participants will make multiple visits to the clinic, and will be contacted by telephone on Day 78 after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Has a primary diagnosis of major depressive disorder (MDD), without psychotic features, according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM 5) criteria, as assessed by a board-certified psychiatrist. MDD should be the principal diagnosis and the condition that best accounts for the clinical presentation. Participants with a secondary diagnosis of generalized anxiety disorder or social anxiety disorder may be included if, in the principal investigator's judgment, such diagnosis will not interfere with participation in the study or with outcome assessments. The diagnostic assessment must include a face-to-face evaluation of the participant using the Mini International Neuropsychiatric Interview (MINI).
2. Has MDD that is resistant to treatment (i.e., TRD), defined as failure to respond to at least 2, but not more than 5, adequate trials of pharmacological treatment in the current episode, as determined using the Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH ATRQ).
3. Qualifies as a candidate for receiving ketamine infusions as a treatment for their depression, in the opinion of the investigator.
4. Is naive to ketamine treatment.
5. Has a Hamilton Depression Rating Scale-17 (HAMD-17) total score of ≥22 at Screening.
6. Is on stable pharmacological treatment for depression (≤50% change in dose) during the last 6 weeks prior to Randomization. Participants who are not currently taking pharmacological treatment for depression may be eligible, with the approval of the medical monitor.

Exclusion Criteria:

1. The participant or any immediate family member has a seizure disorder or a history of seizure disorder, except febrile convulsions.
2. Is currently diagnosed with a personality disorder, dementia, eating disorder, schizophrenia, schizoaffective disorder, or bipolar disorder.
3. Has a history of neurological abnormalities that is judged by the medical monitor to preclude the participant's participation in the study; or brain injury including traumatic injury, perinatal encephalopathy, and postnatal brain damage, blood-brain barrier abnormality, and cavernous angioma.
4. Has a history of cerebral arteriosclerosis.
5. Is currently diagnosed with glaucoma.
6. Is at an imminent risk of suicide per the Columbia - Suicide Severity Rating Scale (C-SSRS) (score of 5) or per the investigator's clinical judgment.
7. Has uncontrolled hypertension or a systolic blood pressure of >150 millimeter of mercury (mm Hg) or diastolic blood pressure >95 mm Hg at Screening.
8. Has a positive urine test result for drugs of abuse (defined as any illicit drug use) at Screening or Day 1.
9. Has a blood alcohol content of ≥0.06% at Screening, prior to ketamine infusion (Day -5 or Day -1), or Day 1.
10. Is currently diagnosed with abuse of or dependence on alcohol or other drugs (except nicotine). The participant will be allowed to enroll if his/her drug and alcohol abuse/dependence is in full (complete, not partial) sustained (>1 year) remission.
11. Has any contraindication to the administration of ketamine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-15 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Time to Relapse of Depressive Symptoms Postdose as Measured by Montgomery Åsberg Depression Rating Scale (MADRS) Total Score | Baseline up to Day 57
  The MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms. Items are rated on scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).

SECONDARY OUTCOMES:
Cohort 1: Change from Baseline in MADRS Total Score at the End of Each Week of Treatment | Baseline and weekly up to Day 57
  The MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms. Items are rated on scale of 0 to 6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Cohort 1: Change from Baseline in Clinical Global Impression-Severity Scale (CGI-S) Score at the End of Each Week of Treatment | Baseline and weekly up to Day 57
  The CGI-S is a 7-point global assessment that measures the clinician's impression of the severity of a participant's illness. It takes into account all available information, such as patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function. A rating of 1 corresponds to "Normal, not at all ill" and a rating of 7 corresponds to "Among the most extremely ill participants." Higher scores indicate more severe illness.
Cohort 1: Change From Baseline in Quick Inventory of Depressive Symptomatology-16 Item (QIDS-SR16) Total Score at the End of Each Week of Treatment | Baseline and weekly up to Day 57
  The QIDS-SR16 is a 16-item self-report measure of depressive symptom severity derived from the 30-item Inventory of Depressive Symptomatology (IDS). The QIDS-SR16 assesses all the criterion symptom domains designated by the American Psychiatry Association Diagnostic and Statistical Manual of Mental Disorders - 4th edition (DSM-IV), to diagnose a major depressive episode. QIDS-SR16 assessment has been used to screen for depression and also to measure symptom severity. This scale is also used to distinguish response from remission, as well as to quantify between group treatments effects in open label and randomized controlled trials. The participant is asked to rate the severity and frequency of specific symptoms present over the last 7 days. The QIDS-SR16 total scores range from 0 to 27.
Cohort 1: Percentage of Participants with Treatment-Emergent Adverse Events (TEAEs) | Baseline up to Day 78
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Cohort 1: Percentage of Participants with Treatment-Emergent Adverse Events (TEAEs) that Led to Study Drug Discontinuation | Baseline up to Day 78
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Cohort 1: Percentage of Participants who Meet the Markedly Abnormal Criteria for Vital Signs Measurement at Least Once Postdose | Baseline up to Day 78
  Vital signs will include body temperature (oral measurement), supine blood pressure (after the participant has rested for at least 5 minutes), respiration rate, and pulse (beats per minute [bpm]).
Cohort 1: Percentage of Participants who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Postdose | Baseline up to Day 78
  The percentage of participants with any markedly abnormal standard safety laboratory values collected throughout the study. Safety Laboratory tests include serum chemistry, hematology and urinalysis.
Cohort 1: Percentage of Participants who Meet the Markedly Abnormal Criteria for Safety Electrocardiogram (ECG) Parameters at Least Once Postdose | Baseline up to Day 78
  The percentage of participants who meet markedly abnormal criteria as measured by a standard 12-lead ECG throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda